CLINICAL TRIAL: NCT03368287
Title: Activity Trackers for Monitoring During Rehabilitation After Total Knee Arthroplasty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Lin Jianhao, The clinical professor of arthritis clinic and research center, Peking University People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PUPH20170958
Record Dates: First submitted 2017-11-25; First posted 2017-12-11 (Actual); Last update posted 2017-12-11 (Actual); Status verified 2017-12

CONDITIONS: Total Knee Arthroplasty
Keywords: Total Knee Arthroplasty; steps; rehabilitation; activity tracker

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- activity tracker (Experimental): In this study, Fitbit One, the activity tracker, will be used for every participants to evaluate the daily steps before and after surgery for one year
  Interventions: Device: Fitbit One, the activity tracker

INTERVENTIONS:
Device: Fitbit One, the activity tracker — Activity tracker, Fitbit One, will be used for a week to evaluate the steps of daily life before the surgery and at the time of follow up.

SUMMARY:
This study aims to estimated the change of the steps of daily life of osteoarthritis patients before and in 6 weeks, 3 months, 6 months, 1 year after the total knee arthroplasty (TKA) through a kind of activity tracker: Fitbit ONE.

DETAILED DESCRIPTION:
A total of 100 participants who will receive total knee arthroplasty will be recruited in this study. Fitbit ONE, the activity tracker, will be used for all of them to monitor the daily steps during the rehabilitation, to be exact, before and at 6 weeks, 3 months, 6 months, 1 year after TKA. Moreover, pain score, self reported questionnaire will also be estimated at those time points.

ELIGIBILITY:
Inclusion Criteria:

* Ready to receive single-side TKA

Exclusion Criteria:

* contraindication of surgery
* self-reported diseases that cause lower limb disability (for example, cerebrovascular disease especially stroke)

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-01-01 (Estimated); Primary Completion 2019-01-30 (Estimated); Study Completion 2019-01-31 (Estimated)

PRIMARY OUTCOMES:
The change of steps of daily life | before operation and 6 weeks, 3 months, 6 months, 1 year after operation
  steps

SECONDARY OUTCOMES:
The change of pain score | before operation and 6 weeks, 3 months, 6 months, 1 year after operation
  Visual Analogue Scale of pain is a scale to estimate pain, and its score ranges from 0 to 10. The higher the score is, the more severe pain the patient is feeling.
The change of knee joint symptoms. | before operation and 6 weeks, 3 months, 6 months, 1 year after operation
  The Western Ontario and McMaster Universities Osteoarthritis Index(WOMAC),and its score ranges from 0 to 96. The higher the score is, the more severe symptoms the patient is feeling.

CONTACTS AND LOCATIONS:
Overall Officials: Jianhao Lin, MD, Principal Investigator — arthritic clinic and research center

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Patel S, Park H, Bonato P, Chan L, Rodgers M. A review of wearable sensors and systems with application in rehabilitation. J Neuroeng Rehabil. 2012 Apr 20;9:21. doi: 10.1186/1743-0003-9-21. PMID 22520559
- [Background] Kooiman TJ, Dontje ML, Sprenger SR, Krijnen WP, van der Schans CP, de Groot M. Reliability and validity of ten consumer activity trackers. BMC Sports Sci Med Rehabil. 2015 Oct 12;7:24. doi: 10.1186/s13102-015-0018-5. eCollection 2015. PMID 26464801
- [Background] Cook DJ, Thompson JE, Prinsen SK, Dearani JA, Deschamps C. Functional recovery in the elderly after major surgery: assessment of mobility recovery using wireless technology. Ann Thorac Surg. 2013 Sep;96(3):1057-61. doi: 10.1016/j.athoracsur.2013.05.092. PMID 23992697